CLINICAL TRIAL: NCT05045131
Title: PeAF-Box. A Study to Investigate the Feasibility, Safety and Efficacy of Isolating the Left Atrial Posterior Wall Adjunctive to Pulmonary Vein Isolation as First-line Therapeutical Strategy in Treatment of Persistent Atrial Fibrillation
Brief Title: PeAF-BOX: Feasibility, Safety and Efficacy of PVI + Box Ablation in Persistent Atrial Fibrillation
Acronym: PeAF-BOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: René Husted Worck (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor-Investigator, René Husted Worck, M.D. Consultant in Cardiology and Cardiac Electrophysiology, University Hospital, Gentofte, Copenhagen
Organization: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PeAF-BOX study
Record Dates: First submitted 2021-09-06; First posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: The PeAF - Box study is observational and investigates single procedure PVI+PWI. Adding PWI to PVI substantially increases the amount of ablation close to the esophagus raising concerns of the risk of esophageal thermal injury. Accordingly, the study includes a formal analysis of the safety of PVI+PWI in terms of risk of esophageal thermal injury. The study includes 24 participants based on power calculations showing that at least 23 participants were required to illustrate a non-inferior risk of inducing esophageal thermal injury by PVI+PWI compared to relevant recently published data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PVI+PWI, 6 months reassessment procedure, 3 year continued rhythm monitoring (Experimental): Single arm experimental, observational study: All participants receive a single-procedure combined PVI + posterior wall isolation (PVI+PWI), loop recorder implantation, esophagoscopy, a mandated interventional reassessment /reablation procedure at six months and continuous rhythm monitoring for three years
  Interventions: Procedure: Left atrial combined pulmonary vein isolation and posterior wall isolation

INTERVENTIONS:
Procedure: Left atrial combined pulmonary vein isolation and posterior wall isolation
  Other Names: Implantation of a subcutaneous cardiac monitor; Interventional reassessment and ablation (if needed) in the left atrium six months after the index procedure

SUMMARY:
Title: PeAF-Box. Feasibility, Safety and Efficacy of Isolating the Left Atrial Posterior Wall (PWI) added to Pulmonary Vein Isolation (PVI) as First-Line Strategy in Treatment of Persistent Atrial Fibrillation (PeAF)

Design: A prospective, observational, single center, unblinded, clinical study with 3 years of follow-up and two interventional procedures: An index ablation procedure and a reassessment/ reablation procedure after 6 months.

Background: In patients with PeAF the effect of first-line ablation with pulmonary vein isolation (PVI) is smaller than in patients with paroxysmal atrial fibrillation (PAF), where PVI alone is effective in reducing symptoms and increasing quality of life. Adding PWI to PVI is increasingly used despite concerns about safety and efficacy.

Objectives: (1) To use PVI + PWI as first-line ablation-strategy in participants with PeAF and to assess the feasibility of obtaining that goal. (2) To assess the safety of applying this lesion set - in terms of heat-induced injury to the esophagus - using esophagoscopy. 3) To asses arrhythmia burden using continuous monitoring for 3 years after ablation. (4) To assess the durability of the PVI + PWI lesion set by a relook/ reablation procedure after 6 months. (5) To follow the effect of PVI + PWI on participants' quality of life over three years.

Study site: Dept of Cardiology - Electrophysiology Laboratory, Gentofte Hospital, University of Copenhagen.

Study population: 24 patients referred for ablation of PeAF are asked for informed consent for these elements that surpass standard treatment in PeAF: (1) Taking amiodarone for 3 weeks prior to the index procedure to 3 weeks after the procedure, (2) Additional ablation with PWI compared to standard first-line therapy with PVI only. (3) Implantation of an implantable cardiac monitor (ICM), (4) Post-procedure esophagoscopy, (5) Regular clinic visits for 3 years post procedure, (6) Undergoing an interventional relook/ reablation procedure 6 months after the index procedure.

Anticoagulation drugs during the procedure and follow up: To prevent thromboses participants are prescribed periprocedural oral anticoagulant treatment to be continued for shorter or longer/lifelong periods according to the participants' risk of thrombosis (the CHA2DS2-VASC score).

Anti-arrhythmic drugs (AADs): Except from periprocedural amiodarone treatment, no AADs are allowed during the follow-up apart from occurrence of otherwise untreatable arrhythmias.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic persistent atrial fibrillation (EHRA symptom class II or above)
* Prior failed treatment with at last one antiarrhythmic drug (Class I-IV)
* Clinical indication for ablation
* Persistent atrial fibrillation meeting both the following requirements:

  * One or more episodes of atrial fibrillation lasting longer than seven days, regardless of mode of termination
  * Estimated cumulated time in PeAF more than 3 months and less than 36 months

Exclusion Criteria:

* Contraindication for ablation
* Predominantly PAF phenotype
* Valvular Heart disease
* Previous ablation in heart
* Previous heart surgery (including valve surgery and coronary artery bypass grafting - CABG)
* Documented atrial flutter or other arrhythmia requiring ablation besides PVI
* Greatly enlarged left atrium on Trans thoracic Echocardiography (TTE ; diameter > 52 mm in males and diameter > 47 mm in females)
* LVEF < 35%
* Implanted pacemaker or defibrillator
* Presence of intramural thombus, tumor or other abnormality precluding catheter introduction
* Pregnancy
* Intolerance to Amiodarone
* Unstable angina pectoris
* Myocardial infarction within 3 months of inclusion
* History of blood clotting or bleeding anomalies
* Malignant disease (non metastatic skin cancer excluded)
* Severe obesity (Mody mass index > 35 kg/m^2)
* Active systemic infection
* Renal insufficiency (serum creatinine > 150 mmoles/liter)
* Psychiatric illness
* Substance abuse
* Participation in other clinical trials

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-03-17 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2020-11-14 (Actual)

PRIMARY OUTCOMES:
The safety of single procedure PVI + PWI | Esophagoscopy is carried out at least 20 hours and less than 48 hours after the index ablation procedure
  Defined as the incidence of inflammation or other injury to the esophagus detected under mandated esophagoscopy on the day after PVI + PWI with radiofrequency ablation. The endoscopy is carried out, assessed and electronically stored by a board-certified gastroenterologist. Metric: n/N in %.

SECONDARY OUTCOMES:
Feasibility of a first-procedure PVI + PWI strategy | The data are available immediately after the end of the index PVI + PWI procedure
  Defined as the ability to achieve complete bidirectional isolation of the left atrial posterior wall as well as all pulmonary veins at a reasonable cost in terms of procedure-, ablation and fluoroscopy times and total patient radiation exposure. Electrical isolation is assessed by visual inspection of electrocardiograms and classical electrophysiological pacing- and sensing maneuvers in the left atrium.
Temperature in the esophagus during radiofrequency ablation | The data are available immediately after the end of the index PVI + PWI procedure
  Defined as the maximum temperature measured in degrees Celsius with one decimal and evaluated for each individual ablation during point-by-point ablations to achieve PVI + PWI. Metric: Degrees Celsius.
Durability of the PVI + PWI lesion set | The data are available immediately after the end of the six months reassessment procedure
  Defined as the proportions of pulmonary veins and left atrial posterior walls remaining durably isolated when controlled at the six months reassessment procedure. Electrical isolation is assessed by visual inspection of electrocardiograms and classical electrophysiological pacing- and sensing maneuvers in the left atrium. Metric: n/N in %.
AF recurrence short term | The data are available 180 days after the index procedure
  Defined as the proportion of participants with recurring atrial fibrillation of at least 2 minutes duration and the time to the first recurrence detected during continuous rhythm monitoring by the implanted loop recorder in the time frame of 90 days from end blanking period to 180 days post index procedure (time of scheduled reassessment procedure). Metric: n/N in %.
AF burden short term | The data are available 180 days after the index procedure
  Defined as cumulated time in atrial fibrillation (minutes) divided by the total number of minutes in the 90 days observation period between end blanking period and time of scheduled reassessment procedure. Metric: min/min in %.
AF recurrence long term | The data are available 1080 days after the index procedure
  Defined as the proportion of participants with recurring atrial fibrillation of at least 2 minutes duration and the time to the first recurrence detected during continuous rhythm monitoring by the implanted loop recorder in the time frame between the reassessment / reablation procedure at 180 days and full three years (1080 days) observation time after the index procedure. Metric n/N in %.
AF burden long term | The data are available 1080 days after the index procedure
  Defined as cumulated time in atrial fibrillation (minutes) divided by the total number of minutes in the 900 days observation period between the 6 months reassessment/ reablation procedure and full three years observation time (1080 days). Moreover, AF burden is calculated every 3 to 6 months during the entire follow - up period. Metric: min./min. in %
Long term efficacy PVI + PWI | The data are available 1080 days after the index procedure
  Defined as incidence of anti arrhythmic drug therapy and repeat ablations between the the reassessment procedure at 180 days and end follow-up at 1080 days. Metric: number of patients and specification of drug
Effect on quality of life by PVI + PWI | Data are available from recruitment to end of follow-up at 3 years
  Defined as self reported scores obtained by repeat answering of the Atrial Fibrillation Effect on Quality of Life (AFEQT) score system. The questionnaire is administered every three to six months to coincide with clinic visits and calculation of AF burden. Metric: range [0-100]

OTHER OUTCOMES:
Time to PVI | Data available immediately after index procedure
  Time from index procedure start until all (or all isolatable) pulmonary veins are electrically isolated at index procedure. Metric: Min.
Time to PVI + PWI | Data available immediately after index procedure
  Time from index procedure start until all (or all isolatable) pulmonary veins and posterior walls are electrically isolated at index procedure. Metric: Min.
Total procedure time | Data available immediately after index procedure
  Time from index procedure start until all catheters are removed from the veins. Metric: Min.
Ablation time PVI | Data available immediately after index procedure
  Cumulated time of radiofrequency (RF) energy delivery required to achieve PVI during index procedure. Metric: min.
Ablation time PVI + PWI | Data available immediately after index procedure
  Cumulated time of RF delivery required to achieve PVI + PWI during index procedure. Metric: min.
Fluoroscopy time PVI | Data available immediately after index procedure
  Cumulated X-ray delivery time from start procedure until PVI achieved during index procedure. Metric: min.
Fluoroscopy time PVI + PWI | Data available immediately after index procedure
  Cumulated X-ray delivery time from start procedure until all catheters removed from the veins in index procedure. Metric: min.
Fluoroscopy dose PVI | Data available immediately after index procedure
  Cumulated X-ray dose to the participant from start procedure until PVI achieved during index procedure. Metric: Gy x cm^2
Fluoroscopy dose PVI + PWI | Data available immediately after index procedure
  Cumulated X-ray dose to the participant from start procedure until all catheters removed from the veins in index procedure. Metric: Gy x cm^2
Index procedure vascular access complications | Data available one month after completion of the index procedure
  The number of participants developing a complication related to vascular access in the right groin. Metric: n/N in %
Index procedure tamponade/ effusions | Data available one day after completion of the index procedure
  The number of participants developing symptoms and signs of pericardial effusion during or after the procedure. Metric: n/N in %
Left atrial volume | Data available after completion of the reassessment procedure
  The left atrial volume before the index procedure and before the reassessment procedure after 6 months. Estimated with 1) Contrast-CT scan of left atrium, 2) Echo - measured left atrial volume and 3) Left atrial volume estimated by electroanatomical mapping (Carto ®, Biosense Webster.Inc). Metric: ml.
Left Ventricular Ejection Fraction (LVEF) | Data available 1 year after the index procedure
  The left ventricular systolic function estimated by LVEF before the index procedure, before the reassessment procedure after 6 months and at 1 year follow-up. Metric: %

CONTACTS AND LOCATIONS:
Overall Officials: René H Worck, MD, Principal Investigator — Herlev-Gentofte Hospital, UCPH

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Worck R, Sorensen SK, Johannessen A, Ruwald MH, Hansen ML, Haugdal M, Hansen J. Posterior wall isolation in persistent atrial fibrillation. Long-term outcomes of a repeat procedure strategy. J Interv Card Electrophysiol. 2023 Jun;66(4):971-979. doi: 10.1007/s10840-022-01402-x. Epub 2022 Nov 3. PMID 36327059
- [Derived] Worck R, Sorensen SK, Johannessen A, Ruwald M, Haugdal M, Hansen J. Posterior wall isolation in persistent atrial fibrillation feasibility, safety, durability, and efficacy. J Cardiovasc Electrophysiol. 2022 Aug;33(8):1667-1674. doi: 10.1111/jce.15556. Epub 2022 May 31. PMID 35598313

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT05045131/Prot_SAP_000.pdf